CLINICAL TRIAL: NCT01050712
Title: Inhaled Carbon Monoxide in Patients With Post-Operative Ileus Following Colon Resection.
Brief Title: Study of Inhaling Carbon Monoxide to Treat Patients With Intestinal Paralysis After Colon Surgery.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: According to retired PI, resident graduated and next resident never carried it to fruition.
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Paul Belliveau, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POICO-B
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Ileus
MeSH Terms: conditions — Ileus | interventions — apoptosis-induced regulator protein

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbon Monoxide (Experimental)
  Interventions: Drug: Inhaled Carbon Monoxide
- Synthetic Air (Placebo Comparator)
  Interventions: Drug: Synthetic Air

INTERVENTIONS:
Drug: Inhaled Carbon Monoxide — Concentration of Carbon Monoxide to be inhaled by patients will be determined in a safety trial performed in healthy volunteers prior to the commencement of this trial. Patients randomized to received inhaled carbon monoxide will receive this concentration by cushioned face mask for one hour prior to colon resection and for one hour after colon resection
  Arms: Carbon Monoxide
Drug: Synthetic Air — Patients randomized to this intervention will receive this gas via cushioned face mask for one hour prior to colon resection and for one hour after colon resection
  Arms: Synthetic Air

SUMMARY:
Post operative ileus (POI), a temporary paralysis of the intestines, is a serious health care problem. It normally occurs in all patients after surgery to the abdomen but in some cases can result in serious complications. The objective of this study is to determine if inhaling very low doses of carbon monoxide (CO) before and after colon surgery will shorten the duration of normal POI and/or prevent the development of POI complications in patients undergoing colon surgery.

A preliminary study will be conducted in six healthy volunteers to monitor for blood levels and adverse effects that occur at 3 different doses of inhaled CO to establish a safe dose for patients in the main trial. For the main trial, patients requiring surgery to their colon will be assigned randomly to receive one hour treatments of either CO or oxygen by face mask before and after their operation. Length of normal POI and occurrence of POI complications will be compared between the two groups. Side effects that occur from inhaling CO or oxygen will also be recorded.

We hypothesize that inhaling CO before and after colon surgery will shorten the length of normal POI and decrease the occurrence of POI complications with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age > 18 years.
* Women must be using acceptable contraceptives, post-menopausal or surgically sterile.
* No prior smoking history.
* BMI between 16 and 30 inclusive.
* No significant abnormalities on history, physical examination or laboratory parameters.

Exclusion Criteria:

* Exposure to any carbon monoxide source during the 48 hours prior to the study day or occupational exposure to CO.
* Significant disease or disorder (as explained in Study B).
* Complete bowel obstruction.
* Intra-abdominal inflammation (diverticulitis, inflammatory bowel disease, colitis).
* Retroperitoneal hematomas.
* Known GI motility disorder.
* Underlying lung disease such as pneumonia, asthma or COPD.
* Sepsis.
* Planned pregnancy, already pregnant or breastfeeding.
* Electrolyte disturbance (hypokalemia, hypomagnesemia, hyponatremia).
* Significant opioid and laxative use 4 weeks prior to surgery.
* Anti-inflammatory use 2 days prior to surgery.
* Drugs such as antacids, Coumadin, amitriptyline, chlorpromazine.
* Baseline oxygen saturation <92% on room air.
* Baseline blood level of COHb >2%.
* Baseline hemoglobin <90 g/dL.
* Participation in another clinical trial within 2 months prior to study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Duration of post operative ileus (radiologic) | 1 week
Incidence of pathological post operative ileus | 1 week
Duration of post operative ileus (clinical) | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Belliveau, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada